CLINICAL TRIAL: NCT07218744
Title: An Open-Label Study Assessing the Mass Balance, Pharmacokinetics, and Metabolite Profiles of a Single Oral Dose of [14C]-INCB123667 in Healthy Male Participants
Brief Title: Study Assessing the Mass Balance, Pharmacokinetics, and Metabolite Profiles of a Single Oral Dose of [14C]-INCB123667 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB123667-103
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: INCB123667

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: INCB123667 (Experimental): Participants will be administered INCB123667 tablet orally, followed approximately 10 minutes later by an oral dose solution of radiolabeled INCB123667.
  Interventions: Drug: INCB123667

INTERVENTIONS:
Drug: INCB123667 — INCB123667 will be administered orally as a tablet dose, followed approximately 10 minutes later by an oral dose solution of radiolabeled INCB123667.

SUMMARY:
This study will assess the mass balance, pharmacokinetics, and metabolite profiles of a single oral dose of [14C] INCB123667 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Healthy males age 18 to 55 years, inclusive, at the time of signing the ICF.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive, at the time of screening.
* No clinically significant findings in screening evaluations (eg, clinical, laboratory, vital signs, ECG). Tests with results that fail eligibility requirements may be repeated once during screening if the investigator believes the results to be in error.
* Ability to swallow and retain oral medication.

Exclusion Criteria:

* History of clinically significant respiratory, renal, GI, endocrine, hematopoietic, psychiatric, and/or neurological disease.
* History of cardiovascular, cerebrovascular, peripheral vascular, or thrombotic disease or uncontrolled hypertension (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg at screening, confirmed by repeat testing).
* Presence of a malabsorption syndrome (eg, Crohn's disease or chronic pancreatitis) that could possibly affect drug absorption.
* Current or recent (≤ 6 months of screening), clinically significant gastrointestinal disease or surgery or any history of GI surgery (including cholecystectomy, excluding appendectomy and uncomplicated hernia repair) that is anticipated to affect the absorption of the study drug.
* Any major surgery within 6 months (≤ 6 months) of screening.
* Donation of blood to a blood bank or participation in a clinical study (except a screening visit) within 4 weeks of screening (within 2 weeks for donation of plasma only).
* Positive test for HBV, HCV, or HIV. Participants whose HBV results are compatible with prior immunization or immunity due to infection may be included at the discretion of the investigator.
* History of significant alcohol use within 3 months of screening, defined as regular alcohol consumption > 21 units per week for males (1 unit = 0.5 pint of beer or a 25-mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type).
* Positive urine or breath test result for ethanol or positive urine or serum screen for drugs of abuse that are not otherwise explained by permitted concomitant medications or diet.
* Current treatment or treatments within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug on Day 1 with another investigational medication, or current enrollment in another investigational drug study.
* Participation in more than 3 radiolabeled drug studies in the last 12 months (previous study in which exposures are known to the investigator to be at least 4 months prior to check-in [Day -1]; previous studies in which exposures are not known to the investigator to be at least 6 months prior to check-in [Day -1]).
* Exposure to significant diagnostic or therapeutic radiation (eg, serial x-ray, computed tomography scan, barium meal) or employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.
* Current treatment or treatment within 15 days or 5 half-lives (whichever is longer) before the first dose of study drug with any medications known to be an inducer or potent inhibitor of CYP3A4, BCRP, or P-gp (refer to the Certara Drug Interaction Database Program for prohibited medications).
* History of tobacco- or nicotine-containing product use within 1 month of screening. However, use of nicotine-containing products that is equivalent to ≤ 2 cigarettes per week may be permitted at the discretion of the investigator.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2025-11-13 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Total Recovery (Urine + Feces) of the Administered Radioactivity | Approximately 2 weeks
  Radioactivity in urine and feces was reported as the percentage of the administered radioactivity excreted.
Percentage of total radioactive dose in Plasma, Urinary and Fecal Excretion | Up to approximately 2 months
  To characterize the metabolic profile and identify circulating and excreted metabolites of INCB123667 following administration of a single oral dose of INCB123667 followed by an oral dose solution of [14C]-INCB123667 using liquid chromatography with mass spectral detection.

SECONDARY OUTCOMES:
PK for plasma INCB123667: Cmax | Up to approximately 2 months
  Defined as the maximum plasma concentration.
PK for plasma INCB123667: tmax | Up to approximately 2 months
  Defined as the time to reach maximum concentration.
PK for plasma INCB123667: AUClast | Up to approximately 2 months
  Defined as area under the concentration-time profile from time zero to time of the last quantifiable concentration (Clast).
PK for plasma INCB123667: AUCinf | Up to approximately 2 months
  Defined as area under the concentration-time profile extrapolated to time of infinity.
PK for plasma INCB123667: t½ | Up to approximately 2 months
  Defined as terminal-phase half-life.
PK for plasma INCB123667: CL/F | Up to approximately 2 months
  Defined as apparent clearance.
PK for plasma INCB123667: Vz/F | Up to approximately 2 months
  Defined as apparent volume of distribution.
PK for whole blood and plasma total radioactivity: Cmax | Up to approximately 2 months
  Defined as the maximum plasma concentration.
PK for whole blood and plasma total radioactivity: tmax | Up to approximately 2 months
  Defined as the time to reach maximum concentration.
PK for whole blood and plasma total radioactivity: t½ | Up to approximately 2 months
  Defined as terminal-phase half-life.
PK for whole blood and plasma total radioactivity: AUClast | Up to approximately 2 months
  Defined as area under the concentration-time profile from time zero to time of the last quantifiable concentration (Clast).
PK for whole blood and plasma total radioactivity: AUCinf | Up to approximately 2 months
  Defined as area under the concentration-time profile extrapolated to time of infinity.
Treatment Emergent Adverse Events (TEAEs) | Up to approximately 2 months
  Adverse events reported for the first time or worsening of a pre-existing event, occurring after study treatment administration.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (1):
- Fortrea Clinical Research Unit Ltd Labcorp Clinical Research Unit Limited Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Assessing the Mass Balance, Pharmacokinetics, and Metabolite Profiles of a Single Oral Dose of [14C]-INCB123667 in Healthy Male Participants — https://incyteclinicaltrials.com/studies/nct07218744